CLINICAL TRIAL: NCT04757636
Title: A Phase 3, Multicentre, Double-masked, Randomised Study to Evaluate the Efficacy and Safety of Intravitreal OPT-302 in Combination With Aflibercept, Compared With Aflibercept Alone, in Participants With nAMD
Brief Title: OPT-302 With Aflibercept in Neovascular Age-related Macular Degeneration (nAMD)
Acronym: COAST
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The primary endpoint was not achieved in the study.
Sponsor: Opthea Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPT-302-1005
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Results first posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-06

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: nAMD; wet AMD; Wet Macular Degeneration; Macular Degeneration; Eye Diseases; Retinal Diseases; Retinal Degeneration
MeSH Terms: conditions — Wet Macular Degeneration; Macular Degeneration; Eye Diseases; Retinal Diseases; Retinal Degeneration | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 2.0 mg aflibercept with Standard Dosing 2.0 mg OPT-302 (Experimental): 2.0 mg aflibercept intravitreal injection administered at 4-weekly intervals for three treatments, and then at 8-weekly intervals.
  2.0 mg OPT-302 intravitreal injection administered at 4-weekly intervals.
  Interventions: Biological: 2.0 mg OPT-302; Biological: 2.0 aflibercept
- 2.0 mg aflibercept with Extended Dosing 2.0 mg OPT-302 (Experimental): 2.0 mg aflibercept intravitreal injection administered at 4-weekly intervals for three treatments, and then at 8-weekly intervals.
  2.0 mg OPT-302 intravitreal injection administered at 4-weekly intervals for three treatments, and then at 8-weekly intervals, with sham intravitreal injection administered at visits when OPT-302 is not.
  Interventions: Biological: 2.0 mg OPT-302; Biological: 2.0 aflibercept
- 2.0 mg aflibercept with sham (Sham Comparator): 2.0 mg aflibercept intravitreal injection administered at 4-weekly intervals for three treatments, and then at 8-weekly intervals.
  Sham intravitreal injection administered at 4-weekly intervals.
  Interventions: Biological: 2.0 aflibercept; Procedure: Sham

INTERVENTIONS:
Biological: 2.0 mg OPT-302 — intravitreal injection
  Arms: 2.0 mg aflibercept with Extended Dosing 2.0 mg OPT-302; 2.0 mg aflibercept with Standard Dosing 2.0 mg OPT-302
Biological: 2.0 aflibercept — intravitreal injection
Procedure: Sham — intravitreal injection
  Arms: 2.0 mg aflibercept with sham

SUMMARY:
A 2-year phase 3, multicentre, randomised, parallel-group, sham-controlled, double-masked study. Primary efficacy will be determined at Week 52.

ELIGIBILITY:
Inclusion Criteria:

* Active subfoveal CNV lesion or juxtafoveal CNV lesion with foveal involvement that is secondary to AMD in the Study Eye.
* An ETDRS BCVA score between 60 and 25 (inclusive) letters in the Study Eye.

Main Exclusion Criteria:

* Any previous treatment for neovascular AMD.
* Clinically significant ocular disorders (other than neovascular AMD), which may interfere with assessment of BCVA, assessment of safety, or fundus imaging.
* Any current (or history of a) social, psychological, or medical condition that precludes enrolment into the study.

  * Additional inclusion/exclusion criteria apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 998 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (179):
- United States (60):
  - COAST Investigational Site, Phoenix, Arizona
  - COAST Investigational Site, Arcadia, California
  - COAST Investigational Site, Huntington Beach, California
  - COAST Investigational Site, Redlands, California
  - COAST Investigational Site, Sacramento, California
  - COAST Investigational Site, Danbury, Connecticut
  - COAST Investigational Site, Altamonte Springs, Florida
  - COAST Investigational Site, Boynton Beach, Florida
  - COAST Investigational Site, Coral Springs, Florida
  - COAST Investigational Site, Melbourne, Florida
  - COAST Investigational Site, Orlando, Florida
  - COAST Investigational Site, Plantation, Florida
  - COAST Investigational Site, Sarasota, Florida
  - COAST Investigational Site, St. Petersburg, Florida
  - COAST Investigational Site, Stuart, Florida
  - COAST Investigational Site, Winter Haven, Florida
  - COAST Investigational Site, Marietta, Georgia
  - COAST Investigational Site, ‘Aiea, Hawaii
  - COAST Investigational Site, Chicago, Illinois
  - COAST Investigational Site, Springfield, Illinois
  - COAST Investigational Site, Urbana, Illinois
  - COAST Investigational Site, New Albany, Indiana
  - COAST Investigational Site, Lenexa, Kansas
  - COAST Investigational Site, Prairie Village, Kansas
  - COAST Investigational Site, West Monroe, Louisiana
  - COAST Investigational Site, Hagerstown, Maryland
  - COAST Investigational Site, Owings Mills, Maryland
  - COAST Investigational Site, Boston, Massachusetts
  - COAST Investigational Site, Worcester, Massachusetts
  - COAST Investigational Site, Jackson, Mississippi
  - COAST Investigational Site, Independence, Missouri
  - COAST Investigational Site, St Louis, Missouri
  - COAST Investigational Site, Edison, New Jersey
  - COAST Investigational Site, Albuquerque, New Mexico
  - COAST Investigational site, Shirley, New York
  - COAST Investigational Site, Asheville, North Carolina
  - COAST Investigational Site, Wilmington, North Carolina
  - COAST Investigational Site, Winston-Salem, North Carolina
  - COAST Investigational Site, Cincinnati, Ohio
  - COAST Investigational Site, Dayton, Ohio
  - COAST Investigational Site, Oklahoma City, Oklahoma
  - COAST Investigational Site, Springfield, Oregon
  - COAST Investigational Site, Kingston, Pennsylvania
  - COAST Investigational Site, Philadelphia, Pennsylvania
  - COAST Investigational Site, Greenville, South Carolina
  - COAST Investigational Site, West Columbia, South Carolina
  - COAST Investigational Site, Rapid City, South Dakota
  - COAST Investigational Site, Germantown, Tennessee
  - COAST Investigational Site, Knoxville, Tennessee
  - COAST Investigational Site, Abilene, Texas
  - COAST Investigational Site, Austin, Texas
  - COAST Investigational Site, Burleson, Texas
  - COAST Investigational Site, Conroe, Texas
  - COAST Investigational Site, Dallas, Texas
  - COAST Investigational Site, Plano, Texas
  - COAST Investigational Site, Round Rock, Texas
  - COAST Investigational Site, Fairfax, Virginia
  - COAST Investigational Site, Bellevue, Washington
  - COAST Investigational Site, Spokane, Washington
  - COAST Investigational Site, Morgantown, West Virginia
- Argentina (4):
  - COAST Investigational Site, Rosario, Santa Fe Province
  - COAST Investigational Site, Rosario, Sante Fe
  - COAST Investigational Site, Ciudad Autonoma de Buenos Aire
  - COAST Investigational Site, Mendoza
- Australia (6):
  - COAST Investigational Site, Liverpool, New South Wales
  - COAST Investigational Site, Parramatta, New South Wales
  - COAST Investigational Site, Strathfield, New South Wales
  - COAST Investigational Site, Adelaide, South Australia
  - COAST Investigational Site, East Melbourne, Victoria
  - COAST Investigational Site, Rowville, Victoria
- COAST Investigational Site, Graz, Austria
- Brazil (3):
  - COAST Investigational Site, Belo Horizonte, Minas Gerais
  - COAST Investigational Site, Porto Alegre, Rio Grande do Sul
  - COAST Investigational Site, São Paulo
- Bulgaria (2):
  - COAST Investigational Site, Sofia
  - COAST Investigational Site, Stara Zagora
- Canada (3):
  - COAST Investigational Site, Brampton, Ontario
  - COAST Investigational Site, North York, Ontario
  - COAST Investigational Site, Ottawa, Ontario
- Colombia (7):
  - COAST Investigational Site, Medellín, Antioquia
  - COAST Investigational Site, Bogotá, Cundinamarca
  - COAST Investigational Site, Cali, Valle del Cauca Department
  - COAST Investigational Site, Barranquilla
  - COAST Investigational Site, Bogotá
  - COAST Investigational Site, Cali
  - COAST Investigational Site, Medellín
- Croatia (3):
  - COAST Investigational Site, Osijek
  - COAST Investigational Site, Split
  - COAST Investigational Site, Zagreb
- Czechia (4):
  - COAST Investigational Site, Hradec Králové, Cech Republic
  - COAST Investigational Site, Brno
  - COAST Investigational Site, Prague
  - COAST Investigational Site, Praha 4-Krc
- COAST Investigational Site, Roskilde, Denmark
- COAST Investigational Site, Tallinn, Estonia
- France (4):
  - COAST Investigational Site, Lyon, Rhone
  - COAST Investigational Site, Poitiers, Vienne
  - COAST Investigational Site, Dijon
  - COAST Investigational Site, Paris
- Germany (4):
  - COAST Investigational Site, Tübingen, Baden Wu
  - COAST Investigational Site, Cologne, North Rhine-Westphalia
  - COAST Investigational Site, Mainz, Rhineland-Palatinate
  - COAST Investigational Site, Berlin
- Greece (4):
  - COAST Investigational Site, Athens
  - COAST Investigational Site, Heraklion
  - COAST Investigational Site, Larissa
  - COAST Investigational Site, Thessaloniki
- Hungary (5):
  - COAST Investigational Site, Budapest
  - COAST Investigational Site, Debrecen
  - COAST Investigational Site, Nyíregyháza
  - COAST Investigational Site, Pécs
  - COAST Investigational Site, Zalaegerszeg
- India (6):
  - COAST Investigational Site, Hyderabad, Andhra Pradesh
  - COAST Investigational Site, Ranchi, Jharkhand
  - COAST Investigational Site, Mysore, Karnataka
  - COAST Investigational Site, Nashik, Maharashtra
  - COAST Investigational Site, Bhubaneswar, Odisha
  - COAST Investigational Site, Madurai, Tamil Nadu
- Israel (5):
  - COAST Investigational Site, Afula
  - COAST Investigational Site, Haifa
  - COAST Investigational Site, Jerusalem
  - COAST Investigational Site, Rehovot
  - COAST Investigational Site, Tel Aviv
- Italy (7):
  - COAST Investigational Site, Ancona, Perugia
  - COAST Investigational Site, Florence
  - COAST Investigational Site, Milan
  - COAST Investigational Site, Pisa
  - COAST Investigational Site, Roma
  - COAST Investigational Site, Rome
  - COAST Investigational Site, Rozzano
- COAST Investigational Site, Riga, Latvia
- Lithuania (3):
  - COAST Investigational Site, Kaunas
  - COAST Investigational Site, Klaipėda
  - COAST Investigational Site, Vilnius
- Netherlands (3):
  - COAST Investigational Site, Nijmegen
  - COAST Investigational Site, Rotterdam
  - COAST Investigational Site, Tilburg
- Philippines (5):
  - COAST Investigational Site, Santo Tomas, Batangas
  - COAST Investigational Site, Makati
  - COAST Investigational Site, Makati City
  - COAST Investigational Site, Pasig
  - COAST Investigational Site, Quezon City
- Poland (7):
  - COAST Investigational Site, Bielsko-Biala
  - COAST Investigational Site, Bydgoszcz
  - COAST Investigational Site, Bytom
  - COAST Investigational Site, Lodz
  - COAST Investigational Site, Lublin
  - COAST Investigational Site, Olsztyn
  - COAST Investigational Site, Poznan
- COAST Investigational Site, Arecibo, Puerto Rico
- Slovakia (4):
  - COAST Investigational Site, Bratislava
  - COAST Investigational Site, Trebišov
  - COAST Investigational Site, Trenčín
  - COAST Investigational Site, Žilina
- South Korea (5):
  - COAST Investigational Site, Seongnam-si, Gyeonggi-do
  - COAST Investigational Site, Suwon, Gyeonggi-do
  - COAST Investigational Site, Busan
  - COAST Investigational Site, Seoul
  - COAST Investigational Site, Soeul
- Spain (7):
  - COAST Investigational Site, Badalona, Barcelona
  - COAST Investigational Site, Majadahonda, Madrid
  - COAST Investigational Site, Oviedo, Principality of Asturias
  - COAST Investigational Site, Barcelona
  - COAST Investigational Site, Madrid
  - COAST Investigational Site, Valencia
  - COAST Investigational Site, Zaragoza
- Taiwan (4):
  - COAST Investigational Site, Kaohsiung City
  - COAST Investigational Site, Taichung
  - COAST Investigational Site, Taipei
  - COAST Investigational Site, Taoyuan
- United Kingdom (9):
  - COAST Investigational Site, Plymouth, Devon
  - COAST Investigational Site, Westcliff-on-Sea, Essex
  - COAST Investigational Site, Manchester, Greater Manchester
  - COAST Investigational Site, Liverpool, Merseyside
  - COAST Investigational Site, Gorleston-on-Sea, Norfolk
  - COAST Investigational Site, Frimley, Surrey
  - COAST Investigational Site, Sunderland, Tyne and Wear
  - COAST Investigational Site, Leeds, West Yorkshire
  - COAST Investigational Site, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants 50 years or older with active subfoveal CNV lesion or juxtafoveal CNV lesion with foveal involvement that is secondary to AMD in the study eye with an ETDRS BCVA score between 60 and 25 (inclusive) letters in the study eye.
Pre-assignment Details: Participants who met all inclusion criteria and none of the exclusion criteria were enrolled in the study.
  2 subjects (in the 2.0 mg aflibercept with sham arm) were enrolled, but never treated.
Groups:
- 2.0 mg Aflibercept With Standard Dosing 2.0 mg OPT-302: 2.0 mg aflibercept intravitreal injection (0.05mL) followed by 2.0 mg OPT-302 intravitreal injection (0.05mL) administered into the study eye at 4-weekly intervals for three treatments, and then at 8-weekly intervals through Week 96, with OPT-302 administered alone at visits when aflibercept was not.
  2.0 mg OPT-302: intravitreal injection
  2.0 aflibercept: intravitreal injection
- 2.0 mg Aflibercept With Extended Dosing 2.0 mg OPT-302: 2.0 mg aflibercept intravitreal injection (0.05mL) followed by 2.0 mg OPT-302 intravitreal injection (0.05mL) administered into the study eye at 4-weekly intervals for three treatments, and then at 8-weekly intervals through Week 96, with sham intravitreal injection administered alone into the study eye at the alternating visits when aflibercept and OPT-302 were not administered.
  2.0 mg OPT-302: intravitreal injection
  2.0 aflibercept: intravitreal injection
  Sham: intravitreal injection
- 2.0 mg Aflibercept With Sham: 2.0 mg aflibercept intravitreal injection (0.05mL) followed by sham intravitreal injection administered into the study eye at 4-weekly intervals for three treatments, and then at 8-weekly intervals through Week 96, with sham intravitreal injection administered alone at visits when aflibercept was not.
  2.0 aflibercept: intravitreal injection
  Sham: intravitreal injection
Period: Overall Study
Arm/Group | 2.0 mg Aflibercept With Standard Dosing 2.0 mg OPT-302 | 2.0 mg Aflibercept With Extended Dosing 2.0 mg OPT-302 | 2.0 mg Aflibercept With Sham
Started (The number of participants randomized into the study) | 333 | 330 | 335
Treated (The number of participants randomized and treated) | 333 | 330 | 333
Completed Week 52 Visit | 300 | 305 | 308
Completed (The number of participants that completed Week 100) | 172 | 173 | 172
Not Completed | 161 | 157 | 163
Not completed — Adverse Event | 25 | 8 | 11
Not completed — Death | 9 | 12 | 6
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 6 | 7
Not completed — Physician Decision | 1 | 3 | 4
Not completed — Withdrawal by Subject | 20 | 23 | 18
Not completed — Discontinued Study Treatment at or prior to Week 52 | 0 | 1 | 0
Not completed — Study Terminated by Sponsor | 103 | 104 | 114
Not completed — Sponsor Decision | 0 | 0 | 1
Not completed — Randomized in Error | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (mITT) dataset comprised all randomised participants with at least one dose of study medication. Participants were analysed according to the study medication to which they were randomised for all efficacy analyses.
  Data from 3 participants at a single site (all randomised to the Aflibercept + Sham arm) were excluded from all analyses based on study site noncompliance with potentially signficant impact to reliability of data.
Groups:
- 2.0 mg Aflibercept With Extended Dosing 2.0 mg OPT-302: 2.0 mg aflibercept intravitreal injection (0.05mL) followed by 2.0 mg OPT-302 intravitreal injection (0.05mL) administered into the study eye at 4-weekly intervals for 3 treatments, and then at 8-weekly intervals through Week 96, with sham intravitreal injection administered alone into the study eye at the alternating visits when aflibercept and OPT-302 were not administered.
  2.0 mg OPT-302: intravitreal injection
  2.0 aflibercept: intravitreal injection
  Sham: intravitreal injection
- 2.0 mg Aflibercept With Sham: 2.0 mg aflibercept intravitreal injection (0.05mL) followed by sham intravitreal injection administered into the study eye at 4-weekly intervals for 3 treatments, and then at 8-weekly intervals through Week 96, with sham intravitreal injection administered alone at visits when aflibercept was not.
  2.0 aflibercept: intravitreal injection
  Sham: intravitreal injection
- Total: Total of all reporting groups
Arm/Group | 2.0 mg Aflibercept With Standard Dosing 2.0 mg OPT-302 | 2.0 mg Aflibercept With Extended Dosing 2.0 mg OPT-302 | 2.0 mg Aflibercept With Sham | Total
Number analyzed (Participants) | 333 | 330 | 330 | 993
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 32 | 34 | 105
  >=65 years | 294 | 298 | 296 | 888
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.3 (7.80) | 74.9 (7.97) | 75.2 (8.28) | 74.8 (8.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 183 | 184 | 557
  Male | 143 | 147 | 146 | 436
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity is only captured in the United States
  Participants
    Hispanic or Latino | 4 | 2 | 6 | 12
    Not Hispanic or Latino | 83 | 81 | 77 | 241
    Unknown or Not Reported | 246 | 247 | 247 | 740
Race (NIH/OMB) [Count of Participants; unit: Participants] — A participant can be considered in more than one race category
  Participants
    American Indian or Alaska Native | 3 | 9 | 6 | 18
    Asian | 29 | 25 | 29 | 83
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 1 | 0 | 0 | 1
    White | 288 | 287 | 281 | 856
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 12 | 9 | 14 | 35
Early Treatment Retinopathy Study (ETDRS) Best-Corrected Visual Acuity (BCVA) Letters [Mean (Standard Deviation); unit: letters read] — The Early Treatment Retinopathy Study (ETDRS) Best-Corrected Visual Acuity (BCVA) letter score at baseline in the study eye.
  letters read | 52.8 (9.04) | 52.3 (9.63) | 52.4 (9.65) | 52.5 (9.44)
Choroidal Neovascularisation (CNV) Area by Fluorescein Angiography (FA) [Mean (Standard Deviation); unit: mm^2] — The Choroidal Neovascularisation (CNV) Area by Fluorescein Angiography (FA) at baseline.
  mm^2 | 6.16 (3.277) | 6.47 (3.137) | 6.54 (3.185) | 6.39 (3.199)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Early Treatment Retinopathy Study (ETDRS) Best-corrected Visual Acuity (BCVA) Letters
Description: To determine the efficacy of intravitreal 2.0 mg OPT-302 when administered in combination with intravitreal 2.0 mg aflibercept, in participants with neovascular age-related macular degeneration (nAMD), in terms of change in ETDRS BCVA letter score in the study eye from Baseline to Week 52. The primary analysis presented used mixed model for repeated measures in the overall population. (A positive outcome measure means an improvement in ETDRS BCVA letter score from baseline; a negative outcome measure means a deterioration in ETDRS BCVA letter score from baseline)
Time Frame: Baseline to Week 52
Population: Modified Intent-to-Treat (mITT) analysis set - comprised all randomised participants with at least one dose of study medication. Participants were analysed according to the study medication to which they were randomised for all efficacy analyses.
Measure: Least Squares Mean (Standard Error); unit: Letters read
Arm/Group | 2.0 mg Aflibercept With Standard Dosing 2.0 mg OPT-302 | 2.0 mg Aflibercept With Extended Dosing 2.0 mg OPT-302 | 2.0 mg Aflibercept With Sham
Number analyzed (Participants) | 333 | 330 | 330
Letters read | 13.48 (0.729) | 12.82 (0.728) | 13.66 (0.728)
Statistical Analysis 1: Comparison: 2.0 mg Aflibercept With Standard Dosing 2.0 mg OPT-302 vs 2.0 mg Aflibercept With Sham; Test type: Superiority; p = 0.861409, MMRM; Least Squares Mean Difference = -0.18, 95% CI 2-sided [-2.20 to 1.84], Standard Error of Mean 1.030
Statistical Analysis 2: Comparison: 2.0 mg Aflibercept With Extended Dosing 2.0 mg OPT-302 vs 2.0 mg Aflibercept With Sham; Test type: Superiority; p = 0.416264, MMRM; Least Squares Mean Difference = -0.84, 95% CI 2-sided [-2.86 to 1.18], Standard Error of Mean 1.029

2. Secondary Outcome: Proportion of Participants Gaining 15 or More ETDRS BCVA Letters
Description: To determine the effects of intravitreal 2.0 mg OPT-302 when administered in combination with intravitreal 2.0 mg aflibercept, in participants with neovascular age-related macular degeneration (nAMD), in terms of proportion of participants gaining 15 or more letters in ETDRS BCVA in the study eye from Baseline to Week 52. The secondary analysis presented used multiple imputation analysis assuming missing at random in the overall population.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- 2.0 mg Aflibercept With Extended Dosing 2.0 mg OPT-302: 2.0 mg aflibercept intravitreal injection (0.05mL) followed by 2.0 mg OPT-302 intravitreal injection (0.05mL) administered into the study eye at 4-weekly intervals for 3 treatments, and then at 8-weekly intervals through Week 96, with sham intravitreal injection administered into the study eye alone at the alternating visits when aflibercept and OPT-302 were not administered.
  2.0 mg OPT-302: intravitreal injection
  2.0 aflibercept: intravitreal injection
  Sham: intravitreal injection
Arm/Group | 2.0 mg Aflibercept With Standard Dosing 2.0 mg OPT-302 | 2.0 mg Aflibercept With Extended Dosing 2.0 mg OPT-302 | 2.0 mg Aflibercept With Sham
Number analyzed (Participants) | 307 | 298 | 303
Participants | 167 | 156 | 162
Statistical Analysis 1: Comparison: 2.0 mg Aflibercept With Standard Dosing 2.0 mg OPT-302 vs 2.0 mg Aflibercept With Sham; Test type: Superiority; p = 0.981348, Mantel Haenszel; Risk Difference (RD) = 0.1, 95% CI 2-sided [-7.5 to 7.7] — The rate/rate differences are estimated and compared by aggregating the MH estimates adjusted for the Baseline BCVA category and baseline lesion type read by independent reading center on each of the 100 multiple imputed datasets using Rubin's rule
Statistical Analysis 2: Comparison: 2.0 mg Aflibercept With Extended Dosing 2.0 mg OPT-302 vs 2.0 mg Aflibercept With Sham; Test type: Superiority; p = 0.856000, Mantel Haenszel; Risk Difference (RD) = -0.7, 95% CI 2-sided [-8.5 to 7.0] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Proportion of Participants Gaining 10 or More ETDRS BCVA Letters
Description: To determine the effects of intravitreal 2.0 mg OPT-302 when administered in combination with intravitreal 2.0 mg aflibercept, in participants with neovascular age-related macular degeneration (nAMD), in terms of proportion of participants gaining 10 or more letters in ETDRS BCVA in the study eye from Baseline to Week 52. The secondary analysis presented used multiple imputation analysis assuming missing at random in the overall population.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 2.0 mg Aflibercept With Standard Dosing 2.0 mg OPT-302 | 2.0 mg Aflibercept With Extended Dosing 2.0 mg OPT-302 | 2.0 mg Aflibercept With Sham
Number analyzed (Participants) | 307 | 298 | 303
Participants | 204 | 197 | 204
Statistical Analysis 1: Comparison: 2.0 mg Aflibercept With Standard Dosing 2.0 mg OPT-302 vs 2.0 mg Aflibercept With Sham; Test type: Superiority; p = 0.655104, Mantel Haenszel; Risk Difference (RD) = -1.7, 95% CI 2-sided [-8.9 to 5.6] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: 2.0 mg Aflibercept With Extended Dosing 2.0 mg OPT-302 vs 2.0 mg Aflibercept With Sham; Test type: Superiority; p = 0.821257, Mantel Haenszel; Risk Difference (RD) = -0.8, 95% CI 2-sided [-8.2 to 6.5] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Change in Choroidal Neovascularisation (CNV) Area by Fluorescein Angiography (FA)
Description: To determine the effects of intravitreal 2.0 mg OPT-302 when administered in combination with intravitreal 2.0 mg aflibercept, in participants with neovascular age-related macular degeneration (nAMD), in terms of change in CNV area as measured by FA in the study eye from Baseline to Week 52. The secondary analysis presented used mixed model for repeated measures in the overall population.
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm^2
Arm/Group | 2.0 mg Aflibercept With Standard Dosing 2.0 mg OPT-302 | 2.0 mg Aflibercept With Extended Dosing 2.0 mg OPT-302 | 2.0 mg Aflibercept With Sham
Number analyzed (Participants) | 290 | 279 | 281
mm^2 | -4.91 (0.165) | -4.92 (0.166) | -4.61 (0.166)
Statistical Analysis 1: Comparison: 2.0 mg Aflibercept With Standard Dosing 2.0 mg OPT-302 vs 2.0 mg Aflibercept With Sham; Test type: Superiority; p = 0.199828, MMRM; Least Squares Mean Difference = -0.30, 95% CI 2-sided [-0.76 to 0.16], Standard Error of Mean 0.234
Statistical Analysis 2: Comparison: 2.0 mg Aflibercept With Extended Dosing 2.0 mg OPT-302 vs 2.0 mg Aflibercept With Sham; Test type: Superiority; p = 0.188725, MMRM; Least Squares Mean Difference = -0.31, 95% CI 2-sided [-0.77 to 0.15], Standard Error of Mean 0.235

5. Secondary Outcome: Proportion of Participants With Absence of Both Sub-retinal Fluid and Intra-retinal Cysts by SD-OCT
Description: To determine the effects of intravitreal 2.0 mg OPT-302 when administered in combination with intravitreal 2.0 mg aflibercept, in participants with neovascular age-related macular degeneration (nAMD), in terms of proportion of participants with absence of both sub-retinal fluid and intra-retinal cysts by SD-OCT in the study eye at Week 52. The secondary analysis presented used multiple imputation analysis assuming missing at random in the overall population.
Time Frame: at Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- 2.0 mg Aflibercept With Extended Dosing 2.0 mg OPT-302: 2.0 mg aflibercept intravitreal injection (0.05mL) followed by 2.0 mg OPT-302 intravitreal injection (0.05mL) administered into the study eye at 4-weekly intervals for 3 treatments, and then at 8-weekly intervals through Week 96, with sham intravitreal injection administered alone into the study at the alternating visits when aflibercept and OPT-302 were not administered.
  2.0 mg OPT-302: intravitreal injection
  2.0 aflibercept: intravitreal injection
  Sham: intravitreal injection
Arm/Group | 2.0 mg Aflibercept With Standard Dosing 2.0 mg OPT-302 | 2.0 mg Aflibercept With Extended Dosing 2.0 mg OPT-302 | 2.0 mg Aflibercept With Sham
Number analyzed (Participants) | 306 | 297 | 301
Participants | 30 | 32 | 29
Statistical Analysis 1: Comparison: 2.0 mg Aflibercept With Standard Dosing 2.0 mg OPT-302 vs 2.0 mg Aflibercept With Sham; Test type: Superiority; p = 0.847810, Mantel Haenszel; Risk Difference (RD) = -0.5, 95% CI 2-sided [-5.6 to 4.6] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: 2.0 mg Aflibercept With Extended Dosing 2.0 mg OPT-302 vs 2.0 mg Aflibercept With Sham; Test type: Superiority; p = 0.718699, Mantel Haenszel; Risk Difference (RD) = 0.9, 95% CI 2-sided [-4.2 to 6.1] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: From Baseline to Week 100
Description: The safety dataset comprised all participants in the mITT dataset (all randomised participants with at least one dose of study medication). Participants were analysed according to the study medication received for all safety analyses. For Other (Not Including Serious) Adverse Events (AEs), non-serious AEs with a frequency greater than 5% within at least one arm are reported; the Total Affected is the total number of participants experiencing at least one non-serious TEAE during the study.
Arm/Group | 2.0 mg Aflibercept With Standard Dosing 2.0 mg OPT-302 | 2.0 mg Aflibercept With Extended Dosing 2.0 mg OPT-302 | 2.0 mg Aflibercept With Sham
All-Cause Mortality (participants affected / at risk) | 9/333 | 12/330 | 6/330
Serious Adverse Events (participants affected / at risk) | 71/333 | 61/330 | 68/330
Other Adverse Events (participants affected / at risk) | 288/333 | 290/330 | 282/330
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.0 mg Aflibercept With Standard Dosing 2.0 mg OPT-302 (N=333) | 2.0 mg Aflibercept With Extended Dosing 2.0 mg OPT-302 (N=330) | 2.0 mg Aflibercept With Sham (N=330)
Visual acuity reduced (Eye disorders) | 2 (2) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 2 (2) | 0 (0)
Cataract nuclear (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract subcapsular (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Lenticular opacities (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 1 (1) — Includes 1 non-study eye event in the Control arm
Retinal haemorrhage (Eye disorders) | 0 (0) | 2 (2) | 2 (2)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Rhegmatogenous retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 2 (2) — Includes 1 non-study eye event in the Extended Dosing arm and 1 non-study eye event in the Control arm
Endophthalmitis (Infections and infestations) | 3 (3) | 0 (0) | 2 (2)
Cataract traumatic (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (3) | 2 (2) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 4 (4) | 4 (4)
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (3) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Degenerative multivalvular disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (2) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Ulcer haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 3 (3)
Pneumonia (Infections and infestations) | 7 (9) | 4 (4) | 7 (7)
Sepsis (Infections and infestations) | 3 (3) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (2) | 1 (1)
Complicated appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Focal peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex hepatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (3)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Aortic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Invasive breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Sarcoma uterus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0)
Encephalitis autoimmune (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Essential tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attach (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vertebrobasilar stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Bladder tamponade (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.0 mg Aflibercept With Standard Dosing 2.0 mg OPT-302 (N=333) | 2.0 mg Aflibercept With Extended Dosing 2.0 mg OPT-302 (N=330) | 2.0 mg Aflibercept With Sham (N=330)
Cataract (Eye disorders) | 83 (87) | 62 (67) | 47 (48) — Includes 24(24) / 21(23) /18(18) participants(events) with non-study eye events in the Standard/Extended/Control arms, respectively
Vitreous detachment (Eye disorders) | 18 (18) | 9 (9) | 6 (7)
Conjunctival haemorrhage (Eye disorders) | 17 (20) | 24 (30) | 13 (15)
Visual acuity reduced (Eye disorders) | 17 (19) | 6 (8) | 13 (20)
Eye pain (Eye disorders) | 16 (34) | 17 (31) | 9 (25)
Retinal degeneration (Eye disorders) | 8 (9) | 13 (13) | 17 (18)
Intraocular pressure increased (Investigations) | 32 (61) | 31 (47) | 11 (17)
Neovascular age-related macular degeneration (Eye disorders) | 29 (30) | 27 (27) | 30 (30) — All events reported are in the non-study eye
COVID-19 (Infections and infestations) | 31 (32) | 32 (32) | 35 (35)
Nasopharyngitis (Infections and infestations) | 22 (25) | 23 (28) | 29 (43)
Urinary tract infection (Infections and infestations) | 18 (22) | 25 (30) | 20 (29)
Influenza (Infections and infestations) | 17 (22) | 12 (14) | 17 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 24 (34) | 14 (20) | 19 (25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (29) | 11 (13) | 13 (23)
Headache (Nervous system disorders) | 18 (27) | 19 (34) | 19 (31)
Hypertension (Vascular disorders) | 12 (15) | 12 (14) | 31 (36)

LIMITATIONS AND CAVEATS:
This study was terminated early by the Sponsor because the study did not meet the primary endpoint. Thus, not all participants in this study completed the full duration of treatment.

Due to clinical program termination, data reported beyond the primary endpoint of Week 52 (safety analysis set) were not held to the expected standards for data verification and cleaning and are reported to the best of Sponsor's ability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principles for publication of results of this study will be addressed in clinical trial agreements between Opthea (Sponsor) and the study site, and Opthea and the subcontractors performing the study. Results means any and all information and know-how (whether patentable or not) which is discovered, invented or developed or which arises in the course of or as a result of the conduct of the Study, including any and all improvements to the products being studied.

DOCUMENTS (2):
  • Study Protocol (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/36/NCT04757636/Prot_001.pdf
  • Statistical Analysis Plan (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/36/NCT04757636/SAP_002.pdf